CLINICAL TRIAL: NCT06290388
Title: A Phase 1/2a, Multicenter, Open-label, Dose Escalation and Expansion Study of Intravenously Administered 23ME-01473 in Participants With Advanced Solid Malignancies
Brief Title: Study of 23ME-01473 in Patients With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor cancelled study
Sponsor: 23andMe, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23ME-01473-CLIN-001
Record Dates: First submitted 2024-02-08; First posted 2024-03-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor
Keywords: Cancer; Phase 1; Solid Tumor; Oncology; NK; ULBP6; Immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 (Experimental): Participants will receive escalating doses of 23ME-01473
  Interventions: Drug: 23ME-01473

INTERVENTIONS:
Drug: 23ME-01473 — 23Me-01473 given by intravenous infusion

SUMMARY:
This is a first-in-human open-label study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of 23ME-01473 given by intravenous infusion in participants with advanced solid cancers who have progressed or are intolerant of available standard therapies.

DETAILED DESCRIPTION:
This study includes a dose escalation portion to determine the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D) to evaluate the clinical activity of 23ME-01473 and further evaluate its safety, tolerability, pharmacokinetics, and pharmacodynamics in participants with solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1: Adults ≥ 18 years of age
2. Phase 1: Histologically-diagnosed locally advanced (unresectable), or metastatic carcinoma or sarcoma that has progressed after standard therapy for the specific tumor type.
3. Adults 18+: Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
4. Life expectancy ≥ 12 weeks
5. Phase 1: Participants with evaluable disease are eligible regardless of tumor type, RECIST 1.1 can be used to assess disease progression.

Exclusion Criteria:

1. Females who are pregnant (positive serum pregnancy test within 7 days prior to study drug administration) or breastfeeding.
2. Immune-Related Medical History

   1. Active autoimmune disease that has required systemic disease-modifying or immunosuppressive treatment within the last 2 years
   2. Receipt of systemic immunosuppressive therapy (e.g. steroids) within 4 weeks prior to the start of study drug administration
   3. History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia, non-infectious pneumonia that required steroids, or evidence of active, non-infectious pneumonitis
   4. History of Grade ≥ 3 immune-mediated toxicity
3. Prior allogeneic or autologous bone marrow transplant, or other solid organ transplant
4. History of a positive test for:

   1. Hepatitis C virus (HCV) infection, except for those who have completed curative therapy for HCV and have undetectable HCV RNA
   2. Hepatitis B virus (HBV) infection, except for those who are receiving treatment with HBV-active nucleos(t)ide antiviral therapy at the time of study entry and have undetectable HBV DNA
   3. Human Immunodeficiency Virus (HIV) infection, except those who meet the following criteria: CD4+ T cells ≥ 350 cells/μL, no history of Acquired Immunodeficiency Syndrome (AIDS)-defining opportunistic infections, HIV RNA < 50 copies/mL, and on a stable antiretroviral regimen for at least 3 months
5. Prior anticancer therapy, including chemotherapy, targeted therapy, biological therapy or immune-checkpoint inhibitors within 4 weeks or 5 drug half-lives (whichever is shorter)
6. History of another malignancy in the previous 2 years, unless cured by surgery alone and continuously disease free.
7. Uncontrolled or symptomatic CNS (central nervous system) metastases and/or carcinomatous meningitis
8. Recent history (within 6 months) of serious cardiovascular disease

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Phase 1:Incidence and severity of dose-limiting toxicities (DLTs) | First dose through 21 days post dose
Phase 1: Incidence and severity of adverse events (AEs) | From Screening through 90 days post treatment
Phase 1 Incidence and severity of serious adverse events (SAEs) | From Screening through 90 days post treatment
ORR based on investigator assessment against RECIST 1.1 criteria | From baseline until disease progression (up to 5 years)

SECONDARY OUTCOMES:
Phase 1: Prevalence and incidence of antidrug antibodies (ADA) to 23ME-01473 | From first dose up to 5 days post treatment discontinuation
Phase 1: Objective response rate (ORR) | From baseline until disease progression (up to 5 years)
  ORR based on investigator assessment against RECIST 1.1 criteria
Duration of response (DoR) | From baseline until disease progression (up to 5 years)
  Duration of response based on investigator assessment against RECIST 1.1 criteria
Disease Control Rate (DCR) | From baseline until disease progression (up to 5 years)
  Disease control rate based on investigator assessment against RECIST 1.1 criteria
Progression free survival (PFS) | From baseline until disease progression (up to 5 years)
  Progression free survival based on investigator assessment against RECIST 1.1 criteria
Time of maximum serum concentration (Tmax) following a single dose of 23ME-01473 | [Time Frame: Cycle 1 (21 days, from Cycle 1 Day 1 predose to Cycle 2 Day 1 predose)]
Area under the concentration-time curve from zero to the last measurable concentration (AUClast) following a single dose of 23ME-01473 | [Time Frame: Cycle 1 (21 days, from Cycle 1 Day 1 predose to Cycle 2 Day 1 predose)]
Last measurable serum concentration (Clast) following a single dose of 23ME-01473 | [Time Frame: Cycle 1 (21 days, from Cycle 1 Day 1 predose to Cycle 2 Day 1 predose)]
Area under the concentration-time curve from zero extrapolated to infinity (AUCinf) following a single dose of 23ME-01473 | [Time Frame: Cycle 1 (21 days, from Cycle 1 Day 1 predose to Cycle 2 Day 1 predose)]
Terminal half-life (T1/2) following a single dose of 23ME-01473 | [Time Frame: Cycle 1 (21 days, from Cycle 1 Day 1 predose to Cycle 2 Day 1 predose]
Maximum serum concentration (Cmax) following multiple doses of 23ME-01473 | [Time Frame: Cycle 4 (21 days, from Cycle 4 Day 1 predose to Cycle 5 Day 1 predose)]
Time of maximum serum concentration (Tmax) following multiple doses of 23ME-01473 | [Time Frame: Cycle 4 (21 days, from Cycle 4 Day 1 predose to Cycle 5 Day 1 predose)]
Area under the concentration-time curve from time zero to the end of the dosing interval (AUCtau) following multiple doses of 23ME-01473 | [Time Frame: Cycle 4 (21 days, from Cycle 4 Day 1 predose to Cycle 5 Day 1 predose)]
Serum concentration at the end of the dosing interval (Ctau) following multiple doses of 23ME-01473 | [Time Frame: Cycle 4 (21 days, from Cycle 4 Day 1 predose to Cycle 5 Day 1 predose)]
Terminal half-life (T1/2) following multiple doses of 23ME-01473 | [Time Frame: Cycle 4 (21 days, from Cycle 4 Day 1 predose to Cycle 5 Day 1 predose)]

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Low, M.D,Ph.D, Study Director — 23andMe, Inc.
Locations (3):
- United States (3):
  - START Midwest, Grand Rapids, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - START Center for Cancer Care, San Antonio, Texas